CLINICAL TRIAL: NCT05577364
Title: A Single-arm, Multi-center, Phase Ib/II Study of Selinexor in Combination With R-CHOP Followed by Selinexor Maintenance for Untreated EBV-positive DLBCL Patients (Xplore Trial)
Brief Title: Selinexor in Combination With R-CHOP Followed by Selinexor Maintenance for Untreated EBV-positive DLBCL Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); Antengene Corporation (Industry)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-534-01
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: EBV-Positive Diffuse Large B-Cell Lymphoma, Nos
Keywords: untreated, EBV-positive diffuse large B-cell lymphoma
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — selinexor; Exportin 1 Protein; R-CHOP protocol; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor in Combination With R-CHOP (Experimental): Patients with untreated EBV-positive diffuse large B-cell lymphoma will receive sequentially higher doses of selinexor in combination with R-CHOP regimen from the second cycle of R-CHOP (3 weeks per cycle).The initial dose of selinexor is 40mg qw po.
  After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with selinexor will be conducted.
  Interventions: Drug: Selinexor; Drug: R-CHOP Protocol

INTERVENTIONS:
Drug: Selinexor — Selinexor: 40mg qw po, and 60mg qw po (phase Ib); RP2D (II study);
  Selinexor is added from the second cycle of R-CHOP regimen.
  Other Names: exportin 1 (XPO1) inhibitor
Drug: R-CHOP Protocol — Rituximab: 375mg/m2 iv.drip D1;
  Cyclophosphamide: 750mg/m2 iv.drip D1;
  Doxorubicin: 50mg/m2 iv.drip D1;
  Vincristine: 1.4g/m2 iv D1;
  Prednisone: 100mg po D1-5;
  Other Names: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone

SUMMARY:
This is a prospective, single-arm, multi-center, phase Ib/II clinical trial to evaluate the safety, tolerability, and efficacy of selinexor in combination with R-CHOP (rituximab, cyclophosphamide, vincristine, doxorubicin, and prednisone) followed by selinexor maintenance for untreated EBV-positive diffuse large B-cell lymphoma (DLBCL) patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, phase Ib/II clinical trial to explore the maximum tolerated dose (MTD) of selinexor when combined with R-CHOP regimen for untreated EBV-positive DLBCL patients.

Phase Ib study:

Selinexor will be given orally at two different doses (40mg qw, and 60mg qw ) and combined with the R-CHOP regimen from the second cycle based on the "3+3" principle.

In the induction therapy period, 6 cycles of R-CHOP regimen and 2 cycles of rituximab in combination with selinexor are planned.

The dose limited toxicity (DLT) will be evaluated after the first cycle of selinexor in combination with R-CHOP.

Phase II study:

The phase II study of selinexor at recommended phase II dose (RP2D) dose level combined with R-CHOP regimen was conducted to explore the efficacy and safety of the combined regimen.

After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with selinexor will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent
2. Age ≥18, ≤70 years, no gender limitation.
3. Histologically confirmed diagnosis of EBV-positive diffuse large B-cell lymphoma (DLBCL) (more than 50% of tumor cells are positive with EBV encoded small RNAs (EBERs) in situ hybridization were considered EBERs positive).
4. Untreated patients, except for the short-time use of prednisone for controlling tumor-induced symptoms (no more than 30mg/d (or other equivalent amounts of other glucocorticoids), no more than 7 days).
5. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma: measurable lesion: Positron emission tomography/computed tomography (PET/CT) or CT and/or MRI, intranodal lesions with long diameter >1.5cm, and short diameter >1.0cm, or extranodal lesions with long diameter > 1.0 cm.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2.
7. Expected survival ≥ 3 months.
8. Adequate function of bone marrow:

   White blood cell ≥3.0×10E9/L, absolute neutrophil count ≥1.5×10E9/L Platelet ≥100×10E9/L (Bone marrow invasive patient≥75×109/L) Hemoglobin≥ 90g/L No granulocyte growth factor, platelet, or red blood cell transfusions were received within 14 days prior to examination.
9. Adequate function of the liver and renal:

   Total bilirubin≤2×upper limit of normal (ULN) (patients with liver invasion or Gilbert syndrome ≤5×ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (patients with liver invasion ≤5×ULN) Serum creatinine ≤1.5×ULN or creatinine clearance rate ≥60 mL/min
10. The patients agree to take effective contraceptive measures during the study period and till 12 months after the last administration of the study treatment.

Exclusion Criteria:

1. EBV-positive DLBCL combined with other types of lymphoma. Transformed DLBCL.
2. EBV-positive DLBCL with central nervous system invasion.
3. The patients had previously received XPO1 inhibitors, such as selinexor and so on.
4. The patients have contraindications to any drug in the combined treatment.
5. The major surgery is performed within 4 weeks before enrollment, except for diagnosis.
6. There are any life-threatening diseases, medical conditions or organ system dysfunction that the investigator believes may affect the safety or compliance of patients.
7. Heart function and disease meet one of the following conditions:

   1. Heart failure with the classification of New York Heart Association heart function of grade II;
   2. A history of unstable angina pectoris;
   3. A history of myocardial infarction within the past 1 years;
   4. Patients with clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. A history of other malignant tumors within the past 5 years (except the cured cervical cancer and basal cell carcinoma of the skin).
9. Patients with active bleeding.
10. Uncontrolled infection exists within 7 days before treatment and parenteral antibiotics, antiviral drugs or antifungal drugs are needed; However, preventive use of these drugs (including parenteral anti-infective drugs) is allowed.
11. Patients with chronic active hepatitis B or active hepatitis C. If the background hepatitis B Surface Antigen (HBsAg) and/or hepatitis B core Antibody (HBcAb) or hepatitis C Virus (HCV) antibody are positive, the further determination for Hepatitis B Virus (HBV) DNA (no more than 2500 copies /mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the assay) can be included. The patients with HBsAg and/or HBcAb positive need to receive anti-HBV drugs.
12. Patients with the infection of human immunodeficiency virus (HIV) and/or acquired Immunodeficiency syndrome.
13. Inability to swallow tablets, presence of malabsorption syndrome, or any other gastrointestinal disease or dysfunction that may affect the absorption of the study drug.
14. Pregnant and lactating women, and subjects of childbearing age who do not want to use contraception.
15. Mentally ill persons or persons unable to obtain informed consent.
16. The investigators think that the patient is not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | The first cycle of selinexor in combination with R-CHOP regimen (21 days)
  To identify the MDT
Recommended Phase II Dose (RP2D) | The first cycle of selinexor in combination with R-CHOP regimen (21 days)
  To identify the RP2D
Complete response rate (CRR) | Up to 24 weeks.
  To investigate the preliminary antitumor efficacy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From date of the first complete response until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Objective response rate (ORR) | Up to 24 weeks.
  To investigate the preliminary antitumor efficacy
Progression-free survival (PFS) | From date of the first injection until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Overall survival (OS) | From date of the first injection until the date of death from ant cause, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Through study completion, an average of 2 years.
  To identify the incidence of AE and SAE

OTHER OUTCOMES:
The correlation between EBV-DNA level and efficacy indicators, such as CRR, DFS, ORR, PFS, and OS | Through study completion, an average of 2 years.
  To explore the correlation between EBV-DNA level and response
The gene mutations such as DDX3X、TET2、PTPN2 and so on are sequenced by whole genome sequencing. | Through study completion, an average of 2 years.
  To explore the correlations between gene mutations and response and prognosis.
The mRNA and lncRNA alterations are sequenced by transcriptome sequencing. | Through study completion, an average of 2 years.
  To explore the correlations between RNA alterations and response and prognosis.
Immune-related indicators such as LAG-3, PD-1, PD-L1, TIGIF, CTLA-4, and so on are assessed by immunohistochemical (IHC) staining. | Through study completion, an average of 2 years.
  To explore the correlations between immune-related indicators and response and prognosis.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Universitiy Cancer Center, Guangzhou, Guangdong
  - Fudan University Shanghai Cancer Center, Shanghai